CLINICAL TRIAL: NCT03456596
Title: Reducing Disparities in Rural Advanced Cancer Patients and Caregivers
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: VA Office of Research and Development (U.S. Federal Agency); University of South Alabama (Other); Spartanburg Regional Healthcare System (Other)
Responsible Party: Principal Investigator, Marie Anne Bakitas, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: X140522006
Record Dates: First submitted 2017-12-18; First posted 2018-03-07 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-02

CONDITIONS: Cancer
Keywords: CBPR; RE-AIM
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Institution: Community cancer centers implementing ENABLE
  Interventions: Other: ENABLE

INTERVENTIONS:
Other: ENABLE — This is an implementation science study in which an evidence-based early palliative care intervention, ENABLE (Educate, Nurture, Advise, Before Life Ends), is being implemented in rural community cancer centers that did not have a palliative care program.

SUMMARY:
The Purpose of this project is to implement ENABLE (Educate, Nurture, Advise, Before Life Ends) at four community cancer practices that have a high percentage of rural and/or medically-underserved patients diagnosed with advanced cancer and their family caregivers. The ENABLE principal investigator (PI) and the Coordinating Center team are located at the University of Alabama at Birmingham (UAB). Site teams are - Spartanburg SC/Gibbs Cancer Center, Birmingham VA Medical Center, University of South Alabama/Mitchell Cancer Institute, UAB Division of Gynecologic Oncology and UAB Department of Hematology Oncology.

DETAILED DESCRIPTION:
ENABLE is an evidence-based concurrent oncology palliative care model that is ready for implementation. It can overcome the barriers created by rural geography and addresses the often unrecognized and unmet needs of the family caregivers. The EIT is an emerging conceptual model for translating evidence into practice. The central core is the linkage between evidence and stakeholders. Successful implementation results from the interaction of Intervention Program/Policy (ENABLE), Implementation Processes (community-based participatory research methods[CBPR] within a learning collaborative) and the Practical Progress Measures (RE-AIM). On-going consideration of the Multi-level Context is pivotal to successful implementation. This approach has the potential to have a high impact on reducing disparities resulting from the gap between ASCO recommendations and current oncology and palliative care practices in rural patients and families.

The Urgent Need to Improve Rural Palliative and End-of-life Care for Patients and Caregivers According to the 2010 US Census data, nearly 60 million citizens live in rural or non-metropolitan areas; however, less than 10% of the 833 US palliative care programs are located in rural areas (data provided by the Center to Advance Palliative Care Registry). Rural advanced cancer patients are vulnerable and at high risk of experiencing social isolation and disparities in palliative care due to long distances from treatment centers, low population density, and limited clinical expertise (because rural primary care clinicians and hospices programs have relatively few terminally-ill patients.) Rural location is related to less and later hospice use. Hence, most rural cancer patients are unlikely to have access to interdisciplinary team-based palliative and hospice care recommended by ASCO2 and National Comprehensive Cancer Network guidelines. These patients will lack this expertise or be transferred to a distant site for palliation.6 Patients transferred to distant tertiary care settings are at high risk of spending their last days or weeks of life far from home and loved ones. Conversely, rural patients may suffer during their last weeks or days of life without the benefit of state-of-art treatments of pain or other causes of distress. A US palliative care report card identified rural location as high risk for little access to palliative care. By definition, palliative care includes family caregiver support. An estimated million Americans are informal caregivers defined as an unpaid individual who assist someone with functional impairment with activities of their daily living to some degree. Informal caregiving can have deleterious effects on the caregivers' physical and emotional health; a phenomenon referred to as caregiver burden. A recent meta- analysis showed that cancer caregivers in particular, compared to non-caregiver controls, exhibited higher levels of stress and depression, and lower subjective well-being and physical health. ENABLE includes the evidence-based, caregiver-specific COPE (Creativity, Optimism, Planning, Expert information) intervention, developed by McMillan and colleagues. COPE, based in problem-solving education theory, is designed to improve caregivers' creative problem-solving, realistic optimism, reasonable goal-setting, and knowledge/utilization of relevant resources. Compared to usual care, two weeks post-intervention, caregivers in COPE showed improvements in caregiver burden and overall QOL. COPE is the basis of the ACS caregiving guide and has been adapted for caregivers in other diseases.

ELIGIBILITY:
Inclusion Criteria:

• Rural serving community-based cancer centers that do not have a palliative care program

Exclusion Criteria

• none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population is rural community-based cancer centers. According to the 2010 US Census data, nearly 60 million citizens live in rural or non-metropolitan areas;however, less than 10% of the 833 US palliative care programs are located in rural areas. Rural advanced cancer patients are vulnerable and at high risk of experiencing social isolation and disparities in palliative care due to long distances from treatment centers,low population density, and limited clinical expertise. Rural location is related to less and later hospice use.Hence, most rural cancer patients are unlikely to have access to interdisciplinary team-based palliative and hospice care recommended by ASCO and National Comprehensive Cancer Network guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2013-07-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
General Organization Index (GOI) Outcomes Measure | 1 Yr Post Implementation
  The General Organizational Index (GOI) is used to describe the organizational strengths of an organization serving healthcare. The total range of the score would be 12 (lowest - no implementation of good organizational structure) to 60 (full implemented organizational structure). The score is derived from 12 categories which are assigned a score of 1 (no implementation) to 5 (fully implemented); hence a total possible score of 12 - 60.

IPD SHARING:
Plan to Share IPD: No